CLINICAL TRIAL: NCT01245517
Title: The Influence of Dietary Phosphorus Education Program on Nutritional Status and Serum Phosphate Level Among Hemodialysis Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Shwu-Huey Yang, Taipei Medical University, School of Nutrition and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99053
Record Dates: First submitted 2010-11-17; First posted 2010-11-22 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Hyperphosphatemia; Malnutrition
Keywords: hyperphosphatemia or malnutrition
MeSH Terms: conditions — Hyperphosphatemia; Malnutrition | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Phosphorus Education Program (Experimental)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Dietary Phosphorus Education Program

SUMMARY:
Aim:

Dietary Phosphorus Education Program can improve patients' knowledge, attitude and behavior of phosphorus restriction diet to reduce the risk of hyperphosphatemia and malnutrition of hemodialysis patients.

Inclusion criteria:

The criteria of subjects are undergoing regular hemodialysis for longer than 3 months at baseline. Subjects' age range is from 20 to 85 years old. Their baseline serum albumin < 4.0 mg/dL, or serum phosphate > 5.0 mg/dL, are eligible for inclusion.

Subjects will be enrolled into this trial after signed informed consent. We expect to recruit 60 subjects. Patients will be excluded if they had liver cirrhosis, malignant tumor, can't finish all education sessions and/or can't complete dietary records monthly. We will recruit a control group into this trial, they are eligible for inclusion but don't want to participant education sessions.

Intervention protocol:

At baseline, the investigators collect demography and pre-test KAP questionnaires among all subjects. If subjects were illiterate then investigator will conduct face-to-face interview and record their answers. Dietary Phosphorus Education is a 6-month program and be implemented by dietitians and investigators, including education, nutritional counseling and dietary records monthly.

The first month was intensive weekly education sessions, each 20 to 30 minutes. Second and third month were monthly education sessions, each 20 to 30 minutes. There are total 6 sessions in this trial. The last 3 months will follow-up periods, will collect anthropometry data monthly, biochemistry measurements and 3-day dietary records among all subjects. If subjects were illiterate then investigator will conduct face-to-face interview or phone-interview to complete each dietary record. Investigator collect post-test KAP questionnaires, diet behavior questionnaires and satisfaction questionnaires from subjects in the end of the trial,. If subjects are illiterate then investigators interview subjects and record.

This is a 6-months trial and retrospective study to collect anthropometry, biochemical measurements and 3-day dietary records from control subjects monthly.

ELIGIBILITY:
Inclusion Criteria:

* The criteria of subjects are undergoing regular hemodialysis for longer than 3 months at baseline. Subjects' age range is from 20 to 85 years old. Their baseline serum albumin < 4.0 mg/dL, or serum phosphate > 5.0 mg/dL, are eligible for inclusion. Subjects will be enrolled into this trial after signed informed consent. We expect to recruit 60 subjects

Exclusion Criteria:

* Patients will be excluded if they had liver cirrhosis, malignant tumor, can't finish all education sessions and/or can't complete dietary records monthly.
* We will recruit a control group into this trial, they are eligible for inclusion but don't want to participant education sessions

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The difference of biochemistry values including phosphate, calcium-phosphate product, albumin, etc. | first month
The difference of knowledge, attitude and practice (KAP) questionnaire's scores during the study program. | third month

SECONDARY OUTCOMES:
To estimate subjects' protein and calorie intake according to 3-day dietary records. | sixth month

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-Huey Yang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan